CLINICAL TRIAL: NCT05519904
Title: Prevalence of Encephalopathy in Patients With Inflammatory Bowel Diseases.
Acronym: PEIBD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre of Postgraduate Medical Education (Other)
Responsible Party: Sponsor
Other Study IDs: nr 59/2022
Record Dates: First submitted 2022-08-26; First posted 2022-08-29 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2022-08

CONDITIONS: Inflammatory Bowel Diseases; Ulcerative Colitis Chronic; Crohn Disease; Irritable Bowel Syndrome; Encephalopathy
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Irritable Bowel Syndrome; Brain Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Inflammatory bowel diseases (IBD), including Crohn's disease and ulcerative colitis, are characterized by extraintestinal manifestations in approximately 30% of cases. Only 3% of these manifestations are neurological diseases, but they have serious consequences for the patient's health, and often constitute a significant diagnostic problem. Neurological symptoms may precede the appearance of IBD symptoms by up to several years. According to the available literature, symptoms of neurological diseases are more common in men and are usually diagnosed after the diagnosis of IBD, but they are rarely associated with exacerbations of the disease. The most common of these are demyelinating diseases such as multiple sclerosis. The very application of treatment in patients with IBD may also play an important role in the development of neurological diseases of various types and pathogenesis. The use of immunosuppressants and therapy with biological drugs may lead to the impairment of the central nervous system due to changes in the white matter of the brain, a predisposition to opportunistic infections, John Cunningham virus infections and the resulting progressive multifocal leukoencephalopathy (PML). So far, the literature describes the occurrence of many neurological diseases in patients with coexisting IBD, caused by side effects of the treatment itself, cerebral vascular diseases or caused by immune disorders. Cases of Wernicke encephalopathy caused by vitamin B1 deficiency have also been reported. A broad term that defines symptoms of not only neurological diseases is encephalopathy. By definition, it means damage or disease that affects the brain. It occurs when the way the brain works is changed due to a change in the body. These changes cause changes in the psyche, causing confusion and a change in typical behavior. Encephalopathy is not a single disease entity but a disorder with complex pathophysiology. It is a serious disease that, if untreated (or rather its underlying cause), leads to permanent brain damage. Due to the variety of symptoms and their variable severity, the diagnosis of encephalopathy often escapes the team of chronically ill patients. Patients with IBD are such a group - young patients whose severe, incurable disease changes their philosophy of life. The influence of IBD on encephalopathy symptoms has not been evaluated so far. This study is designed to answer the question of whether encephalopathy occurs in people with IBD. By extrapolating the incidence of encephalopathy in people with another immunologically mediated disease, Hashimoto's disease, we hypothesized that such a disorder could also occur in people with IBD. We assume that autoimmune mechanisms underlying the disease will contribute to the etiopathogenesis of the phenomenon, similarly to thyroid disease. Additionally, with increasing incidence in the scientific literature, it is stated that in about 30% of cases, IBD symptoms overlap with functional bowel diseases such as Irritable Bowel Syndrome (IBS), so we plan, in the questionnaire presented to patients, to include questions regarding the coexistence of these disorder as described in the Roman IV Criteria.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Inflammatory Bowel Disease (Ulcerative Colitis, Crohn's Disease)

Exclusion Criteria:

* The study group will exclude people who do not respond to pharmacological treatment, including biological / biomimetic drugs, and will be referred for surgery, as well as people with previously diagnosed neuropsychiatric diseases. In addition, the study will exclude patients with nervous system diseases and liver diseases who are suspected or diagnosed with encephalopathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with inflammatory bowel diseases who within 12 months were:
  * hospitalized at the Department of Gastroenterology in Bielanski Hospital in Warsaw,
  * patients consulted at the Gastroenterology Outpatient Clinic
  * patients reporting for outpatient endoscopic examinations at the Endoscopy Unit Among these people, a group of patients treated with biological or biomimetic drugs will be distinguished, due to the correlation, as indicated in the literature, between the use of anti-TNF drugs and the occurrence of disturbances in the functioning of the nervous system.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of encephalopathy in patients with Inflammatory Bowel Disease | 2-3 Months
  Finding the presence or absence of symptoms of encephalopathy in people with IBD

SECONDARY OUTCOMES:
Number of patients with overlapping symptoms of Inflammatory Bowel Diseases and Irritable Bowel Syndrome | 2-3 Months
  In addition, due to the fact that in about 30% of cases, the overlap of IBD symptoms with functional bowel diseases, such as Irritable Bowel Syndrome (IBS), we are planning presented to patients, include questions regarding the coexistence of these disorders described in the Roman IV Criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Pietrzak, MD, Principal Investigator — Medical Centre of Postgraduate Education
Locations (1):
- Szpital Bielański im. Jerzego Popiełuszki, Warsaw, Masovian Voivodeship, Poland